CLINICAL TRIAL: NCT06171100
Title: Efficacy and Safety of Low-dose Tolvaptan in Treatment of Inpatient Hyponatraemia.
Brief Title: Low-dose Tolvaptan for Inpatient Hyponatraemia.
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GafREC: Endo205
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Hyponatremia; SIADH
Keywords: Tolvaptan
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First dose tolvapatan
  Interventions: Drug: Tolvaptan
- Second dose tolvaptan
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Oral ingestion of low dose Tolvaptan (7.5mg daily) for management of inpatient hyponatraemia for 1st dose Tolvaptan group.
  Oral ingestion of low dose Tolvaptan (7.5mg daily) or standard dose Tolvaptan (15mg daily) for 2nd dose Tolvaptan group.

SUMMARY:
This is a retrospective cohort study to assess the safety and efficacy of low first dose of Tolvaptan and low or standard second dose of Tolvaptan in patients with moderate to severe hyponatraemia associated with SIADH not responding to conservative means of hyponatraemia management.

Patients are treated as part of standard clinical care. There is growing evidence that treating patients with SAIDH induced hyponatraemia using a low dose of Tolvaptan with 7.5mg (below licensed lowest 15mg daily dose). This is the largest study to date and seeks to validate the efficacy and safety or this lower than approved dose of Tolvaptan in patietns who only need a first dose but also in patients who need a second low or srandard dose of Tolvaptan.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Accident & Emergency department or seen as inpatients with moderate to severe hyponatraemia (sNa: <125mmol) associated with SIADH and not responding to conservative measures of hyponatraemia management.
* Patients of all genders aged 18-90 y.o

Exclusion Criteria:

* Pregnant women and patients aged < 18y.o
* Hyponatraemia not associated with SIADH

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital through Accident & Emergency department or those who developed inpatient moderate to severe refractory hyponatraemia associated with SIADH and needed treatment with Tolvaptan.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Response to low dose tolvaptan | Within 30 hours from tolvaptan intake
  Evaluate the efficacy of tolvaptan 7.5mg daily to improve sodium concentration during inpatient hyponatraemia
Safety of low dose tolvaptan | Within 30 hours from tolvaptan intake
  Evaluate the magnitude of sodium increase after an initial 7.5mg Tolvaptan dose

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom